CLINICAL TRIAL: NCT05531084
Title: Safety and Effectiveness of Surgeon-Modified Fenestrated and Branched Endografts in Treating Subjects With Complex Aortic Aneurysms
Brief Title: Safety and Effectiveness of Surgeon-Modified Stent Grafts forTreatment of Complex Aortic Aneurysms
Acronym: Assets
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jesse Manunga, MD (Other)
Collaborators: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor-Investigator, Jesse Manunga, MD, Vascular and Endovascular Surgeon, Minneapolis Heart Institute Foundation
Organization: Minneapolis Heart Institute Foundation (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1861968
Record Dates: First submitted 2022-08-08; First posted 2022-09-07 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Thoracoabdominal Aneurysm; Juxtarenal Aortic Aneurysm; Pararenal Aneurysm; Aortic Aneurysm; Failed Previous Infrarenal Repairs (Failed EVAR)
Keywords: surgeon-modified fenestrated stent grafts
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Intervention Model Description: All participants will receive the same treatment modality (surgeon-modified fenestrated stent grafts).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Thoracoabdominal aortic aneurysm extent I-III (Experimental): Thoracoabdominal aortic aneurysm extent I-III (proximal seal can be from the left carotid artery to directly after the left subclavian artery):
  Interventions: Device: Surgeon-Modified fenestrated stent grafts using Cook Zenith Platform (Zfen, TX2, Alpha Thoracic Endovascular Graft and Zenith Flex)
- Failed EVAR (Experimental): Failed EVAR (defined as type IA endoleak or increase in aneurysm sac size in the setting of proximal seal loss)/juxtarenal/Pararenal/paravisceral/thoracoabdominal aortic aneurysm extent IV-V:
  Interventions: Device: Surgeon-Modified fenestrated stent grafts using Cook Zenith Platform (Zfen, TX2, Alpha Thoracic Endovascular Graft and Zenith Flex)

INTERVENTIONS:
Device: Surgeon-Modified fenestrated stent grafts using Cook Zenith Platform (Zfen, TX2, Alpha Thoracic Endovascular Graft and Zenith Flex) — Depending on the location of the aneurysm, patients with failed EVAR and complex aortic pathology requiring fenestrated and branched endovascular repair will be treated with physician-modified Cook Zenith devices (Zenith Flex, Zenith Fenestrated stent graft (Zfen), Cook Alpha Thoracic Endovascular Graft, Cook dissection TX2), and their associated commercially approved ancillary components.
  Other Names: Cook Zenith Alpha Thoracic Endovascular Graft (P140016); Cook Zenith Fenestrated AAA Endovascular Graft (P020018 S044); Cook Zenith TX2 Dissection Endovascular Graft (P180001); Cook Zenith Flex AAA Bifurcated Main Body (P020018 S055); Atrium iCAST covered Stent (K050814); Gore Viabahn VBX Balloon Expandable Endoprosthesis (P160021)

SUMMARY:
The primary objective of the present study is to evaluate the safety, effectiveness, and clinical outcomes of surgeon-modified fenestrated stent grafts used to treat patients with failed previous infrarenal repairs (failed EVAR) and complex aortic aneurysms (thoracoabdominal, juxtarenal, pararenal, and paravisceral aneurysms).

DETAILED DESCRIPTION:
The study is a prospective, non-randomized evaluation of endovascular repair of patients with failed previous infrarenal repairs (failed EVAR) and complex thoracoabdominal/juxtarenal/pararenal/paravisceral aortic aneurysm repair, including those with penetrating ulcers and aneurysms resulting from aortic dissections, who (1) have anatomy that is not suitable for endovascular repair using grafts currently marketed in the United States, (2) are deemed unsafe to wait the required time necessary for commercial endograft manufacturing, and (3) are at high risk for open surgical repair.

Depending on the location of the aneurysm, patients with failed EVAR and complex aortic pathology requiring fenestrated and branched endovascular repair will be treated with physician-modified Cook Zenith devices (Zenith Flex, Zenith Fenestrated stent graft (Zfen), Cook Alpha Thoracic Endovascular Graft, Cook dissection TX2), and their associated commercially approved ancillary components. Whenever possible, the Zenith fenestrated universal bifurcated device will be used for patients requiring repair down to the iliac arteries. The Gore Excluder Endoprosthesis or the Gore Iliac Branch Endoprosthesis (IBE) will be used whenever the Zenith universal bifurcated device is not available. Safety and effectiveness will be assessed acutely (i.e., treatment success and technical success), at 30 days (i.e., the rate of major adverse events (MAE)), at 6 months, at 12 months, and annually to 5 years (i.e., the proportion of treatment group subjects that achieve and maintain treatment success).

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old
* The subject has one or more of the following:

  1. An aneurysm with a maximum diameter of > 5.5 cm (in men) and 5 cm (in women) or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e, perpendicular to the centerline) measurements 2. Aneurysm with a history of growth > 0.5 cm in 6 months or clinically indicated for repair based on symptoms 3. Symptomatic aneurysm 4. Ruptured aneurysm 6. Failed previous EVAR defined as type IA endoleak or increase in aneurysm sac size in the setting of proximal seal loss 7. Saccular aneurysm deemed by the treating vascular specialist at significant risk for rupture 8. High risk for open surgical repair based on any of the factors below:

  a. Anatomic i. Previous abdominal surgery ii. Previous left-sided thoracotomy (if the proposed open repair would require dissection of the thoracic aorta) iii. Previous aortic surgery b. Physiological high risk For this IDE, physiological risk will be assessed using two systems. First, this study will use the Society for Vascular Surgery (SVS)/American Association for Vascular Surgery (AAVS) medical comorbidity grading system recommended for use by the SVS to describe the severity of medical comorbidities in patients with complex aortic aneurysm disease. However, as the current SVS/AAVS grading system has yet to be validated in prospective studies or in a large cohort of patients treated for aortic disease, the American Association of Anesthesiologists grading system will also be utilized due to its widely adopted use and simplicity although it relies on subjective parameters and lacks specific metrics that affect outcomes.
* American Association of Anesthesiologists grading system: subjects with ASA scores of 3-5 will be considered for study inclusion though final subject approval will be at the discretion of the treating vascular specialist; subjects with ASA scores of 6 will be excluded.
* SVS/AAVS grading system: high risk (8-20% mortality risk) subjects will be considered for study inclusion though final subject approval will be at the discretion of the treating vascular specialist; prohibitive high risk (31-70% mortality risk) subjects will be excluded.

Medical Inclusion Criteria

* American Association of Anesthesiologists (ASA) physical status classification system: subjects with ASA scores of 1-5 will be considered for study inclusion though final subject approval will be at the discretion of the treating vascular specialist; subjects with ASA scores of 6 will be excluded.

SVS/AAVS grading system: low risk (0.12-1% mortality risk), medium risk (1.7-4.9% mortality risk), and high risk (8-20% mortality risk) subjects will be considered for study inclusion though final subject approval will be at the discretion of the treating vascular specialist; prohibitive high risk (31-70% mortality risk) subjects will be excluded.

Anatomical Inclusion Criteria

* Iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices, or accessories, with or without use of a surgical conduit
* Extent of aorta to be treated: infrarenal aortic aneurysms with < 10 mm neck length, juxtarenal or pararenal aneurysms that include 1 or 2 renal arteries; paravisceral and extent IV-V thoracoabdominal aneurysms, Extent I-III thoracoabdominal aneurysm including those patients requiring a carotid-left subclavian bypass in order to achieve, at least, 20 mm of proximal landing zone
* Non-aneurysmal aortic segment proximal to the aneurysm (neck) with a:

  1. Minimum neck length of 20 mm
  2. Diameter in the range of 20 mm - 38 mm
  3. Angle less than 60 degrees relative to the axis of the aneurysm
  4. Angle less than 60 degrees relative to the axis of the suprarenal aorta
* Minimum branch vessel diameter of 5 mm or greater Iliac artery distal fixation site greater than 45 mm in length and diameter in the range of 8 mm to 17 mm

Exclusion Criteria:

* Age: < 18 years old
* Does not meet the above inclusion criteria
* Can be treated in accordance with the instructions for use with a commercially approved and marketed endovascular prosthesis
* Is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site with the exception of percutaneous aortic valve surgery
* Unwilling or unable to comply with the follow-up schedule
* Inability or unwillingness of patient or patient's legally authorized representative to provide informed consent.
* Subject is pregnant or breastfeeding
* Any other circumstance or condition which, at the discretion of the sponsor-investigator, makes the patient unsuitable for inclusion Medical Exclusion Criteria
* Known sensitivities or allergies to the materials of construction of the devices, including but not limited to titanium and PTFE.
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Subject has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned < 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest, or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome, Ehler's Danlos Syndrome) with the exception of patients who have had prior open surgical aortic replacement where a surgical graft would serve as a "landing zone" for the investigational stent-graft Anatomical Exclusion Criteria

  1. Significant occlusive disease, tortuosity, or calcification that would prevent endovascular access
  2. Proximal neck length ≤20 mm
  3. Proximal neck, measured outer wall to outer wall on a sectional image (CT)

     1. For use of Zenith Fenestrated: diameter >32 mm or <18 mm
     2. For use of Zenith Alpha Thoracic: diameter >38 mm or <18 mm (for proximal and distal neck diameter)
     3. Zenith TX2 Dissection Endovascular graft: diameter 38 mm or <18 mm
     4. Zenith Flex AAA endovascular graft: diameter >32 mm or < 18 mm
  4. Proximal neck angulated more than 60 degrees relative to the long axis of the aneurysm
  5. Proximal neck diameter changes over the length of the proximal seal zone >4 mm
  6. Proximal seal site with a circumferential thrombus/atheroma
  7. Iliac artery diameter, measured inner wall to inner wall on a sectional image (CT) <7.0 mm at any point along access length (prior to deployment)
  8. Ipsilateral iliac artery fixation site diameter, measured inner wall on a sectional image (CT) >21 mm at distal fixation site
  9. Iliac artery distal fixation site <10 mm in length
  10. Non-bifurcated segment of any artery to be stented < 15 mm in length
  11. Artery to be stented with a maximum diameter <3 mm or >10 mm at the vessel ostium
  12. Inability to maintain at least one patent hypogastric artery
  13. Bilateral renal artery stenosis >80%
  14. Superior mesenteric artery stenosis >80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Prevention of aortic aneurysm related mortality and all cause mortality post intervention | 5 years
  Primary outcome criteria:
  * Mortality related to primary aortic disease and intervention
  * All-cause mortality post intervention

SECONDARY OUTCOMES:
Issues associated with disease progression, branched instability, endoleak and other disabling complications as evaluated on post-operative follow up and radiographic images. | 5 years
  Secondary outcome criteria (as evidenced on follow up imaging and laboratory tests):
  * Evidence of aortic disease progression (aneurysm growth >/=5 mm)
Endoleak | 5 years
  presence of any endoleak requiring intervention
Target vessels instability resulting in adverse events to the patient | 5 years
  * mesenteric ischemia
  * renal failure
procedure related complication | 5 years
  * stroke
  * Myocardial infarction
  * Paraplegia
Issues associated with device migration and failure | years
  - Device failure (migration >/=10 mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No